CLINICAL TRIAL: NCT00174434
Title: A Phase 1 Study Of Paclitaxel In Combination With SU011248 For Patients With Breast Cancer As First-Line Treatment In The Advanced Disease Setting
Brief Title: Study Of SU011248 In Combination With Paclitaxel In Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181073
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2009-01-27 (Estimated); Status verified 2008-10

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Sunitinib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: SU011248; Drug: Paclitaxel

INTERVENTIONS:
Drug: SU011248 — SU011248 provided as capsules. The starting dose is 25 mg orally, daily in a continuous regimen beginning on day 2. Dose rest for 1 week is allowed. Dose escalation to 37.5 mg po OD is allowed within the constraints of acceptable toxicity parameters. Dosing will continue for 1 year or until disease progression or unacceptable toxicity, whichever comes first.
  Other Names: sunitinib malate, Sutent
Drug: Paclitaxel — Paclitaxel is provided as an intravenous infusion for 1 hour weekly for 3 weeks followed by a 1-week rest. The starting dose is 90 mg/m2. The weekly dose may be decreased to 65 mg/m2 in subsequent cycles based on tolerability. Dosing will continue for 1 year or until maximum benefit, disease progression or unacceptable toxicity, whichever comes first.

SUMMARY:
This study is to evaluate the safety of SU011248 in combination with paclitaxel in patients with metastatic or locally recurrent breast cancer who have not received chemotherapy treatment in the advanced disease setting.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer with evidence of unresectable, locally recurrent or metastatic disease.
* Candidate for treatment with paclitaxel.

Exclusion Criteria:

* Prior chemotherapy in the advanced disease setting.
* HER2 positive disease unless previously treated with trastuzumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Safety of the combination of SU011248 and paclitaxel | 9/05-7/07

SECONDARY OUTCOMES:
Pharmacokinetics of each medication | 9/05-7/07
Objective disease response | 9/05-7/07
Progression-free survival. | 9/05-7/07

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Pfizer Investigational Site, Harvey, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Munster, Indiana
  - Pfizer Investigational Site, New York, New York

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181073&StudyName=Study%20Of%20SU011248%20In%20Combination%20With%20Paclitaxel%20In%20Patients%20With%20Metastatic%20Breast%20Cancer%20%20